CLINICAL TRIAL: NCT06977490
Title: Human Bioequivalence Study of Amphotericin B Liposome for Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sichuan Huiyu Pharmaceutical Co., Ltd (Industry)
Collaborators: Changsha King-eagle Med Technology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JY-BE-AMB-2024-120
Record Dates: First submitted 2025-04-30; First posted 2025-05-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Invasive Fungal Infections; Neutropenic Fever; Visceral Leishmaniasis
MeSH Terms: conditions — Invasive Fungal Infections; Febrile Neutropenia; Leishmaniasis, Visceral | interventions — Amphotericin B; Injections; Long-Term Synaptic Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Amphotericin B Liposome for Injection (Sichuan Huiyu Pharmaceutical Co., Ltd.) (Experimental): * Amphotericin B Liposome for Injection (strength: 50 mg, Sichuan Huiyu Pharmaceutical Co., Ltd.)
  * The test product
  Interventions: Drug: Amphotericin B Liposome for Injection (strength: 50 mg, Sichuan Huiyu Pharmaceutical Co., Ltd.)
- Amphotericin B Liposome for Injection (trade name: Ambisome®) (Experimental): * Amphotericin B Liposome for Injection (trade name: Ambisome®, strength: 50 mg, MAH: Gilead Sciences)
  * The reference product
  Interventions: Drug: Amphotericin B Liposome for Injection (trade name: Ambisome®, strength: 50 mg, MAH: Gilead Sciences)

INTERVENTIONS:
Drug: Amphotericin B Liposome for Injection (strength: 50 mg, Sichuan Huiyu Pharmaceutical Co., Ltd.) — Single intravenous administration of 3.0 mg/kg in each period.
  Other Names: The test product
  Arms: Amphotericin B Liposome for Injection (Sichuan Huiyu Pharmaceutical Co., Ltd.)
Drug: Amphotericin B Liposome for Injection (trade name: Ambisome®, strength: 50 mg, MAH: Gilead Sciences) — Single intravenous administration of 3.0 mg/kg in each period.
  Other Names: The reference product
  Arms: Amphotericin B Liposome for Injection (trade name: Ambisome®)

SUMMARY:
Single-center, randomized, open-label, single-dose, two-treatment, two-period, two-sequence crossover design to evaluate the human bioequivalence of two Amphotericin B Liposome for Injection formulations

DETAILED DESCRIPTION:
To evaluate the human bioequivalence of Amphotericin B Liposome for Injection (strength: 50 mg) provided by Sichuan Huiyu Pharmaceutical Co., Ltd. and Amphotericin B Liposome for Injection (trade name: Ambisome®, strength: 50 mg, MAH: Gilead Sciences) by comparing the differences in the extent and rate of absorption between the two formulations in a healthy Chinese population under a single-center, randomized, open-label, single-dose, two-treatment, two-period, two-sequence crossover design.

ELIGIBILITY:
Inclusion Criteria:

The enrolled participants shall meet all of the following criteria:

1. The study participants must give informed consent before the trial, fully understand the content, process and possible adverse reactions, and voluntarily sign a written informed consent;
2. The study participants can communicate well with the investigators and complete the trial according to protocol;
3. Sex: female or male; age: 18-50 years (inclusive);
4. Body Mass Index (BMI): 19-28 kg/m2 (inclusive), with a minimum weight of 50.0 kg for males and 45.0 kg for females (BMI = Body weight / Height2 [kg/m2]).

Exclusion Criteria:

Study participants meeting one or more of the following criteria will be excluded:

1. Allergic constitution (such as those allergic to two or more drugs or foods [e.g., milk], or pollen), or known history of allergy to the components of the study drug or similar drugs (API: amphotericin B; excipients: hydrogenated soy phosphatidylcholine, cholesterol, distearoylphosphatidylglycerol [sodium salt], alpha tocopherol, sucrose, disodium succinate hexahydrate, hydrochloric acid, and sodium hydroxide); (inquiry)
2. Subjects with the following diseases of clinical significance (including but not limited to diseases related to respiratory system, circulatory system, digestive system, blood system, endocrine system, immune system, skin system, psycho-neurological system, ophthalmology and otorhinolaryngology); (inquiry)
3. Subjects with gastrointestinal, liver and kidney diseases that affect the pharmacokinetics of drugs; (inquiry)
4. Subjects who underwent major surgery within 6 months prior to initial administration, or who planned to undergo surgery during the study; (inquiry)
5. Clinically significant abnormalities in vital signs, physical examination, electrocardiogram and laboratory tests (blood biochemistry, hematology, urinalysis, coagulation); (as determined by the clinical investigator)
6. Subjects with a history of hepatitis B, hepatitis C, AIDS (Acquired Immune Deficiency Syndrome), syphilis and/or abnormalities in one or more of the four tests for infectious diseases with clinical significance; (as determined by the clinical investigator)
7. Blood loss or blood donation of greater than or equal to 400 mL within 3 months prior to initial administration (except for female menstrual period), and/or platelet donation within 2 weeks prior to initial administration; (inquiry)
8. Use of any prescription medicine within 14 days prior to initial administration or use of any over-the-counter medicine, Chinese herbal medicine or health product within 7 days prior to initial administration (except for topical drugs with local effects); (inquiry)
9. Use of azoles (e.g., ketoconazole, miconazole, clotrimazole, fluconazole, etc.), skeletal muscle relaxants, corticosteroids and adrenal cortical hormones, antineoplastic agents, digitonin, flucytosine or other nephrotoxic medications within 28 days prior to initial administration; (inquiry)
10. Subjects who received vaccines or live attenuated vaccines within 4 weeks prior to the administration of the study drug, or who planned to be vaccinated during the trial; (inquiry)
11. Subjects who received medication in any clinical trial or participated in any medical device clinical trial within 3 months prior to initial administration; (inquiry + online screening)
12. A history of drug abuse within 5 years, and/or drug use within 3 months prior to screening, and/or habitual use of any drug (including Chinese herbs) or positive urine drug screening; (inquiry + as determined by the clinical investigator)
13. Subjects who smoked more than 5 cigarettes per day within 3 months prior to screening and/or did not agree to refrain from using any tobacco products during the trial; (inquiry)
14. Regular drinkers within 6 months prior to screening, i.e., subjects who drank more than 14 units of alcohol per week (1 unit = 360 mL of beer with 5% alcohol or 45 mL of spirits with 40% alcohol or 150 mL of wine with 12% alcohol), or subjects who did not agree to stop drinking alcohol 48 h prior to initial administration and during the trial, or test positive for breath alcohol;
15. Subjects who consume excessive amounts of tea, coffee and/or caffeinated beverages (more than 8 cups, 1 cup = 250 mL) per day within 6 months prior to screening, and/or do not agree that tea, coffee and/or caffeinated foods, grapefruit and/or grapefruit juice, and/or products containing opium poppy are prohibited 48 h prior to initial administration and during the trial; (inquiry)
16. Subjects who have a birth plan (including sperm or egg donation) and/or do not agree to take effective contraceptive methods (non-drug during the trial period) from signing informed consent form to 6 months after the final administration; (inquiry)
17. Pregnant or lactating women or subjects with positive pregnancy results; (inquiry, for females only)
18. Subjects who have used oral contraceptives within 30 days prior to initial administration; (inquiry)
19. Use of long-acting estrogen and/or progesterone injections and/or implants within 6 months prior to initial administration; (inquiry, females only)
20. Women of childbearing age who have unprotected sex with their partner within 14 days prior to initial administration; (inquiry, females only)
21. Subjects who cannot tolerate venipuncture or have a history of needle and blood sickness; (inquiry)
22. Subjects who may not be able to complete the study for other reasons or who the investigator considers should not be included.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2025-05-13 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2025-10-07 (Actual)

PRIMARY OUTCOMES:
Cmax | 0 hour before safe dose and 0 hour before formal dose to 1320 hours post formal dose
  90% confidence interval is within the 80.00%-125.00% equivalence margin.
AUC0-t | 0 hour before safe dose and 0 hour before formal dose to 1320 hours post formal dose
  90% confidence interval is within the 80.00%-125.00% equivalence margin.
AUC0-∞ | 0 hour before safe dose and 0 hour before formal dose to 1320 hours post formal dose
  90% confidence interval is within the 80.00%-125.00% equivalence margin.
AUC0-10h | 0 hour before safe dose and 0 hour before formal dose to 1320 hours post formal dose
  90% confidence interval is within the 80.00%-125.00% equivalence margin.
AUC10-last | 0 hour before safe dose and 0 hour before formal dose to 1320 hours post formal dose
  90% confidence interval is within the 80.00%-125.00% equivalence margin.

SECONDARY OUTCOMES:
Tmax | 0 h before safe dose and 0 h before formal dose to 1320 hours post formal dose
  90% confidence intervals will also be investigated as supportive data.
λz | 0 h before safe dose and 0 h before formal dose to 1320 hours post formal dose
  90% confidence intervals will also be investigated as supportive data.
t1/2 | 0 h before safe dose and 0 h before formal dose to 1320 hours post formal dose
  90% confidence intervals will also be investigated as supportive data.
AUC_%Extrap | 0 h before safe dose and 0 h before formal dose to 1320 hours post formal dose
  90% confidence intervals will also be investigated as supportive data.

CONTACTS AND LOCATIONS:
Overall Officials: Qing Wen, Study Director — Jinan Central Hospital
Locations (1):
- Jinan Central Hospital, No.105, Jiefang Road,, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No